CLINICAL TRIAL: NCT00160238
Title: A Double-Blind, Placebo-Controlled, Randomized, Clinical Study of the Effects of Betaserc® 24 mg (1 Tablet b.i.d Over 3 Months) on Vestibular Compensation Following Vestibular Neurotomy in Patients With Disabling Menière's Disease
Brief Title: Effects of Betaserc on Vestibular Compensation in Patients Suffering From Disabling Meniere's Disease and Having Undergone Vestibular Neurotomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S108.4.102
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2006-12-22 (Estimated); Status verified 2006-12

CONDITIONS: Meniere's Disease
Keywords: Meniere's disease; Vestibular neurotomy
MeSH Terms: conditions — Meniere Disease | interventions — Betahistine; BID protein, human

INTERVENTIONS:
Drug: Betahistine 24 mg bid (Betaserc)

SUMMARY:
This study is to compare the effects of Betaserc 24mg and placebo on compensation of postural and locomotor deficits (static and dynamic posturography) after vestibular neurotomy in patients suffering from disabling Menière's disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone vestibular neurotomy for the treatment of disabling Menière's disease and who have confirmed vestibular areflexia

Exclusion Criteria:

* Other peripheral vestibular disease than Menière's disease
* Central vestibular disease
* Neurological disease
* Contraindication to betahistine
* Pregnant or lactating women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2003-01

PRIMARY OUTCOMES:
Patients who have undergone vestibular neurotomy for the treatment of disabling Menière's disease and who have confirmed vestibular areflexia

SECONDARY OUTCOMES:
Other peripheral vestibular disease than Menière's disease;Central vestibular disease; Neurological disease; Contraindication to betahistine; Pregnant or lactating women

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (1):
- Site 1, Marseille, France